CLINICAL TRIAL: NCT06526624
Title: ARTEMIS-009: A Phase 3, Randomized, Controlled, Multi-center, Open-label Study of HS-20093 Versus Active Surveillance As Consolidation Therapy After Chemoradiotherapy in Subjects With Limited-Stage Small Cell Lung Cancer
Brief Title: A Study of HS-20093 vs Active Surveillance in Limited-Stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-20093-302
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Limited-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HS-20093 (Experimental): Patients with LS-SCLC who have not progressed following CRT. Patients in this arm will be administrated HS-20093 intravenously at a dose of 8.0 mg/kg, Q3W continuously until disease progression or until other criteria for discontinuation of treatment are met.
  Interventions: Drug: HS-20093
- Active surveillance (No Intervention): Patients with LS-SCLC who have not progressed following CRT. Patients in this arm will receive active surveillance until disease progression or until other criteria for discontinuation of active surveillance are met.

INTERVENTIONS:
Drug: HS-20093 — Subjects in experimental arm will be given HS-20093 intravenously at a dose of 8.0 mg/kg every 3 weeks, until disease progression or until other criteria for treatment discontinuation are met.
  Arms: HS-20093

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of HS-20093 compared with active surveillance as consolidation therapy after chemoradiotherapy in participants with limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, multi-center, phase III clinical study to evaluate the efficacy and safety of HS-20093 versus active surveillance as consolidation therapy in participants with limited-stage small cell lung cancer (LS-SCLC) who have not progressed after receiving chemoradiotherapy (CRT).

This study consists of an experimental arm and a control arm. The experimental arm will be administered HS-20093, and the control arm will only receive active surveillance. Efficacy and safety were assessed in both arms by follow-up analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed Informed Consent Form.
2. Males or females ≥18 years old.
3. Patients with limited-stage SCLC who are deemed unsuitable for surgery or decline surgery.
4. ECOG performance status of 0-1.
5. Patients who have received CRT and have not progressed.
6. Minimum life expectancy > 12 weeks.
7. Males or Females should be using adequate contraceptive measures throughout the study.
8. Females must not be pregnant at screening or have evidence of non-childbearing potential.

Exclusion Criteria:

1. Patients with mixed SCLC or NSCLC or sarcoma-like carcinoma, or large cell neuroendocrine carcinoma.
2. Patients with extensive-stage SCLC.
3. Disease progression during CRT or before randomization.
4. Received or are receiving the following treatments:

   1. For LS-SCLC, prior treatment with or current use of other chemotherapy regimens other than platinum plus etoposide
   2. Received any other anti-cancer treatment.
   3. Previous or current treatment with B7-H3 target therapy.
   4. Traditional Chinese medicine indicated for tumors within 2 weeks prior to the first dose of study drug.
   5. Major surgery within 4 weeks prior to the first dose of study drug.
5. Interstitial lung disease (ILD)/non-infectious pneumonitis.
6. History of other primary malignancies.
7. Inadequate bone marrow reserve or organ functions.
8. Severe, uncontrolled or active cardiovascular disorders.
9. Severe or uncontrolled diabetes.
10. Serious or poorly controlled hypertension.
11. Severe bleeding symptoms or bleeding tendencies within 1 month prior to randomization.
12. Severe arteriovenous thrombosis occurred within 3 months prior to randomization.
13. Serious infection within 4 weeks prior to randomization.
14. Presence of Grade ≥ 2 toxicities due to prior anti-tumor therapy.
15. Having serious neurological or mental disorders.
16. History of hypersensitivity to any component of HS-200093 or its similar drugs.
17. Participants with any condition that compromises the safety of the participant or interferes with the assessment of the study, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) According to RECIST v1.1 by Independent Review Committee (IRC) | Approximately 6 years
  To assess the efficacy of HS-20093 vs active surveillance in terms of PFS. PFS is defined as the time from randomization until the date of objective disease progression or death, whichever occurred first, based on IRC using RECIST v1.1.
Overall survival (OS) | Approximately 6 years
  To assess the efficacy of HS-20093 vs active surveillance in terms of OS. Overall Survival is defined as the time from the date of randomization to the date of participant's death due to any cause.

SECONDARY OUTCOMES:
PFS at 12 Months (PFS12) or 18 Months (PFS18) According to RECIST v1.1 by IRC | Approximately 6 years.
  PFS12 and PFS18 are defined as the progression-free survival at 12 months and 18 months from the date of randomization, respectively, based on IRC using RECIST v1.1.
ORR According to RECIST v1.1 by IRC | From the date of randomization until the date of disease progression or withdrawal from study, up to approximately 6 years.
  ORR is defined as the percentage of participants with BOR of CR or PR per RECIST v1.1
DCR According to RECIST v1.1 by IRC | From the date of randomization until the date of disease progression or withdrawal from study, approximately 6 years.
  DCR is deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease)
DoR by IRC | From the date of CR, PR until the date of disease progression or death, approximately 6 years.
  DoR only applies to participants whose best overall response is CR or PR. The start date is the date of first documented response of CR or PR, and the end date is defined as the date of the first documented progression or death due to underlying disease.
PFS According to RECIST v1.1 by investigators (INVs) | Approximately 6 years.
  PFS is defined as the time from randomization until the date of objective disease progression or death, whichever occurred first, based on INVs using RECIST v1.1
PFS12 or PFS18 According to RECIST v1.1 by INVs | Approximately 6 years.
  PFS12 and PFS18 are defined as the progression-free survival at 12 months and 18 months from the date of randomization, respectively, based on INVs using RECIST v1.1.
ORR According to RECIST v1.1 by INVs | From the randomization until the date of disease progression or withdrawal from study, up to approximately 6 years.
  ORR is defined as the percentage of participants with BOR of CR or PR per RECIST v1.1 by INVs.
DCR According to RECIST v1.1 by INVs | From the randomization until the date of disease progression or withdrawal from study, up to approximately 6 years.
  DCR is deﬁned as the percentage of patients who have a best overall response (CR, PR, or stable disease).
DoR According to RECIST v1.1 by INVs | From the date of first dose until the date of disease progression or withdrawal from study, up to approximately 6 years.
  DoR is deﬁned as the percentage of patients who have a best overall response (CR, PR, or stable disease).
Proportion of patients alive at 24 months (OS24) or 36 months (OS36) | Approximately 6 years.
  OS24 and OS36 are defined as the proportion of patients alive at 24 months and 36 months from the date of randomization, respectively, based on INVs using RECIST v1.1.
Incidence and severity of treatment-emergent adverse events | From the date of first dose until 90 days after the final dose. A cycle is 21 days.
  Adverse event (assessed according to NCI CTCAE v5.0) is defined as any untoward medical occurrence in a participant without regard to possibility of causal relationship.